CLINICAL TRIAL: NCT00785837
Title: Effects of Hydrotherapy in Pain and Quality of Sleep's Cycles in Preterm Newborn on Neonatal Intensive Care Units
Acronym: hydrotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Luterana do Brasil (Other)
Responsible Party: CARINE MORAES VIGNOCHI, ULBRA - UNIVERSIDADE LUTERANA DO BRASIL
Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: hydrotherapy
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-09

CONDITIONS: Perinatal Care
Keywords: Hydrotherapy; Perinatal Care; Neonatology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Before Hidrotherapy (No Intervention)
- Hidrotherapy (Experimental)
  Interventions: Other: Aquatic Physical Therapy

INTERVENTIONS:
Other: Aquatic Physical Therapy — The Physiotherapy was performed with gentle movements in eight shape, from left to right, in addition to movements of unbundling girdle, light and slow the trunk and extremities posture and body by flexing the organization Wrapping the body.
  Arms: Hidrotherapy

SUMMARY:
Researchers suggest that the protection of the cycles of sleep is essential for neurodevelopment, learning, memory and preservation of brain plasticity to the individual's life. Recent research shows that technical bath promote reduction of crying, anxiety and improves the behavior of newborns.

DETAILED DESCRIPTION:
This was a pilot study assessing the technique in this population. The study was conducted with 8 stable premature infants admitted in the Neonatal Intensive Care Unit (ICU) from Hospital Luterano de Porto Alegre. Physiological and behavioral parameters were assessed by Brazelton's neonatal behavior assessment scale, and the pain was evaluated by NFCS scale. The mean of Brazelton's scale was reduced after the procedures from 5,88 ± 0.35 to 1,38 ± 0.74, p < 0.001. The score in pain assessment scale was reduced from 5,38 ± 0.91 to 0.25 ± 0.46, p < 0.001 after intervention. The study suggests that aquatic physical therapy could be a simple and effective method to reduce pain and stress in premature infants admitted in the neonatal ICU.

ELIGIBILITY:
Inclusion Criteria:

* premature infants with gestational age less than 36 weeks,
* clinically stable, showing behavioral abnormalities such as intolerance to the touch, excessive crying, showing signs of pain in accordance with the scale
* difficulty of NFCS leave the stage of crying and agitation for a period of deep sleep during a period of not less than 60 minutes.

Exclusion Criteria:

* premature medically unstable because of the difficulty of monitoring in liquid medium, with a change in temperature on mechanical ventilation who had an infectious process due to the exacerbation of it in hot water, and syndromic children with congenital facial deformities that impede the use of scale NFCS for evaluation.

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-09 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Physiological and behavioral parameters were assessed by Brazelton's neonatal behavior assessment scale, and the pain was evaluated by NFCS scale. The mean of Brazelton's scale was reduced after the procedures from 5,88 ± 0.35 to 1,38 ± 0.74, p < 0.001. | At two years

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Luterana Do Brasil, Canoas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Vignochi CM, Teixeira PP, Nader SS. Effect of aquatic physical therapy on pain and state of sleep and wakefulness among stable preterm newborns in neonatal intensive care units. Rev Bras Fisioter. 2010 May-Jun;14(3):214-20. English, Portuguese. PMID 20730365